CLINICAL TRIAL: NCT03351322
Title: A Randomized, Double-Blind, Active-controlled, Parallel, Phase II Study to Evaluate Efficacy and Safety of ENERGI-F701 Solution in Female Subjects With Hair Loss
Brief Title: ENERGI-F701 for Female Hair Loss Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Energenesis Biomedical Co., Ltd. (Industry)
Collaborators: A2 Healthcare Taiwan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENERGI-F701-01
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Female Pattern Baldness; Hair Loss; Alopecia
Keywords: Alopecia; Hair Loss; Female Pattern Baldness
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ENERGI-F701 (Experimental): ENERGI-F701, topical application (1 mL) on the scalp of affected area, twice daily for 12 weeks
  Interventions: Drug: ENERGI-F701
- Regaine (Active Comparator): Regaine, topical application (1 mL) on the scalp of affected area, twice daily for 12 weeks
  Interventions: Drug: Regaine

INTERVENTIONS:
Drug: ENERGI-F701 — ENERGI-F701 are applied for treatment of hair loss.
  Arms: ENERGI-F701
Drug: Regaine — Regaine are applied for treatment of hair loss.
  Arms: Regaine

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of ENERGI-F701 Solution in female subjects with hair loss.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged at least 20 years old
2. With hair loss over 100 hairs/day
3. Willing to maintain the same hair style, color, shampoo and hair products used, and approximate hair length starting from signing ICF and throughout the study
4. The subject of childbearing potential must show a negative urine or serum pregnancy test at Screening Visit
5. Have signed the written informed consent form

Exclusion Criteria:

Any subject meeting any of the exclusion criteria will be excluded from study participation.

1. With alopecia areata or cicatricial alopecia
2. With other scalp or hair disorders
3. With prior hair transplant
4. Use wigs or hair weaves
5. Plan to use any other concomitant therapy to treat hair loss, regrowth or volume during the study
6. Have taken any topical or systemic prescription of OTC medications for treating hair loss, hair regrowth and/or hair volume
7. Have used medications known to cause hair thinning, such as Coumadin and anti-depressants/anti-psychotics
8. Have received chemotherapy/cytotoxic agents as well as radiation/laser/surgical therapy of the scalp
9. Have initiated or terminated the use of hormones for birth control or hormone replacement therapy within 6 months. Subject will also be excluded from the study if she plans to initiate or terminate the use of hormones for birth control or hormone replacement therapy during the study.
10. With known or suspected hypersensitivity any ingredients of study product and active control
11. Any hematologic abnormalities.
12. Any serum chemistry abnormalities.
13. Pregnant, lactating, or premenopausal with childbearing potential but not adopting at least one form of birth control.
14. Enrollment in any investigational drug trial
15. With any condition judged by the investigator that entering the trial may be detrimental to the subject

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
The amount of hair loss | Week 12
  Change of the amount of hair loss at Week 12 from baseline.(hair loss is defined as the collection of hairs after combing at the study site)

SECONDARY OUTCOMES:
The amount of hair loss at each post-treatment visit | Week 2, 4, 6, 8, 10
The thickness and density of hair | Week 2, 4, 6, 8, 10, 12
  Change of hair thickness and density measured by phototrichogram at each post-treatment visit
Investigator assessment at each post-treatment visit | Week 2, 4, 6, 8, 10, 12
  The hair loss will be assessed by the investigator using Investigator Photographic Assessment Questionnaire (IPAQ).The change from Baseline in hair growth will be assessed using the following 7-point scale: -3 = greatly decreased, -2 = moderately decreased, -1 = slightly decreased, 0 = no change, +1 = slightly increased, +2 = moderately increased, +3 = greatly increased.
The hair wash/shed hair count at each post-treatment visit | Week 2, 4, 6, 8, 10, 12
  Subjects will collect hairs full day, including after combing and hair-washing. Subjects should turn in these hair collections at each visit. The results will be averaged weekly.
The subject satisfaction | Week 2, 4, 6, 8, 10, 12
  Subject satisfaction evaluated by Women's Androgenic Alopecia Quality of Life Questionnaire (WAA-QOL) at each post-treatment visit from baseline. WAA-QOL is a sixteen-question questionnaire to evaluate subjects' quality of life influenced by hair loss. Each question will be assessed using the following 7-point scale: 0 = not at all, 1 = a little bit, 2 = somewhat, 3 = a good bit, 4 = quite a bit , 5 = very much, 6 = extremely.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided